CLINICAL TRIAL: NCT00194467
Title: Suppression of Oral Shedding of Human Herpesvirus 8 (HHV-8) With Valganciclovir
Brief Title: Suppression of Oral HHV8 Shedding With Valganciclovir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Corey Casper, MD, MPH, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 02-1500-B; VAL041
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Human Herpesvirus 8
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: valganciclovir
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: valganciclovir — 900 mg once a day for 8 weeks
  Other Names: Valcyte
  Arms: 1
Drug: placebo — matching placebo, once a day for 8 weeks
  Arms: 2

SUMMARY:
The purpose of the study is to use valganciclovir to define the role of antiviral therapy in suppression of HHV-8 shedding in HHV-8 seropositive men. Our hypothesis is that valganciclovir will substantially reduce the frequency of detection and amount of HHV-8 in the mouth.

DETAILED DESCRIPTION:
The purpose of the study is to use valganciclovir to define the role of antiviral therapy in suppression of HHV-8 shedding in HHV-8 seropositive men. Our hypothesis is that valganciclovir will substantially reduce the frequency of detection and amount of HHV-8 in the mouth. Such reduction will serve to confirm that the mouth is the site of active HHV-8 replication. If valganciclovir is found to be effective, the findings from this proposal would serve as the basis for a clinical trial with valganciclovir for prevention of Kaposi's Sarcoma (KS) in high-risk HHV-8 seropositive persons.

After informed consent, all subjects will undergo medical history, physical examination and screening laboratory examination. Eligible patients will return to clinic for randomization to receiver either valganciclovir 900 mg qd or placebo. Participants will receive a diary for noting adverse events and concurrent medications. The clinician will instruct the participants on collection of mouth swabs and provide Dacron swabs, vials with PCR media and pre-printed labels. Subjects will be asked to obtain a swab of oral mucosa every morning. Clinic visits every other week will serve to review interim medical history and diaries for adverse events, collect PCR swabs, dispense additional medication and draw safety labs. The study uses a double-blind, randomized placebo design. Therefore, participants will not know whether they will be taking a placebo or active medication at any time during the study. Due to the crossover study design, however, all participants will receive the same amount of placebo and study drug over the duration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* HHV-8 seropositive or previous evidence of HHV-8 shedding
* a frequent shedder of HHV-8
* not receiving any drugs with known anti-HHV-8 activity for study duration
* able to comply with the study protocol
* agree to HIV testing

Exclusion Criteria:

* history of evidence of CMV disease
* hypersensitivity to ganciclovir or valganciclovir
* use of high-dose acyclovir, valacyclovir, famciclovir, ganciclovir, foscarnet, or cidofovir
* neutropenia
* renal insufficiency with serum creatinine greater than 1.5mg.ml or CrCl less than 60
* AST or ALT greater than 5 times upper limit of normal
* concurrent administration of medications which are often associated with severe neutropenia or thrombocytopenia
* concurrent administration of probenecid or didanosine

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The reduction in percent days on which HHV-8 is detected on versus off valganciclovir. The quantitative reduction in the HHV-8 DNA detected by PCR on versus off valganciclovir. | 19 weeks

SECONDARY OUTCOMES:
The frequency of neutropenia, defined as ANC less than 500. The frequency of thrombocytopenia, defined as platelets less than 75,000. | 19 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States